CLINICAL TRIAL: NCT07152067
Title: Stereotactic Focal Radiotherapy as an Alternative Treatment to Active Surveillance for Low and Intermediate Risk Prostate Cancer: a Multicentric Phase-II Randomized Trial
Brief Title: Stereotactic Focal Radiotherapy as an Alternative Treatment to Active Surveillance for Low and Intermediate Risk Prostate Cancer
Acronym: TOPPGUN-RS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, NICKERS Philippe, Clinical Professor, Centre Hospitalier Universitaire de Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/176; B7072025000023 (Registry Identifier: Comité d'Ethique Hospitalo-Facultaire Universitaire de Liège)
Record Dates: First submitted 2025-08-12; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Macroscopic Tumor Visualized at MRI; Tumor Size Allowing Partial Prostate Treatment Volume; CAPRA SCORE ≤5
Keywords: radiosurgery; focal treatment; early prostate cancer; active surveillance; Phase II randomized study; stereotactic radiotherapy; SBRT; quality of life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Patients will be randomized between active surveillance or stereotactic radiation focused on the Index prostatic lesion visualized at MRI exams
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Surveillance (No Intervention): Active surveillance involving MRI, follow-up biopsies and PET PSMA exams
- Focal stereotactic radiation treatment (Experimental): Focal radiation treatment followed by MRI, prostate biopsies and PET PSMA follow up exams
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT to the macroscopic prostate tumor component defined at MRI
  Other Names: Focal stereotactic radiation treatment
  Arms: Focal stereotactic radiation treatment

SUMMARY:
*Rationale : Active surveillance of prostate cancer helps to avoid the morbidity associated with curative radical prostatectomy /radiotherapy in patients with early stage disease. However, at 5 years and 15 years, respectively 35 % and nearly 50 % of patients require rescue interventional treatments. Numerous Phase II trials have reported using focal treatments (focused on the macroscopic tumor only while not involving the whole prostatic gland) in order to reduce the morbidity due to recurrence as well as the high anxiety rates under observation only. Stereotactic radiotherapy (highly focused radiotherapy technic to reduce the risk of side effects) is being proposed in the same way as it does not require any anaesthesia, as opposed to all the other focal methods. The purpose of this trial is to evaluate whether focal stereotactic radiotherapy treatments could reduce the rate of rescue treatments among patients eligible to an active surveillance program at first.

* Major Inclusion Criteria :

  * 1. Early stage prostate adenocarcinoma (CAPRA score ≤ 5)
  * 2. No major urinary problems
  * 3. Active Surveillance possible
* Major Exclusion Criteria :

  * 1. Age at diagnosis < 50 years
  * 8. Androgen-deprivation therapy
  * 9. Any cancer within the last 5 years except skin basocellular carcinoma or any uncontrolled cancer
* Trial : Phase II randomized trial comparing Stereotactic Radiation Therapy focused on the macroscopic tumor or Active Surveillance as the control arm.
* Main objective : to compare the rescue treatment rates between the two arms

DETAILED DESCRIPTION:
The stereotactic radiation therapy procedure involves at first placement of 3-4 fiducial markers, a planning computed tomography (CT) scan as well as a planning MRI, both fused thereafter based on fiducial markers. The delay between fiducial markers placement and planning CT Scan - MRI must be of at least 10 days. SBRT delivers 36.25 Gy in 5 fractions prescribed on the 80% isodose or higher. The fractions are delivered with a CyberKnife device every other day for 2 weeks. If constraints to organs at risk can be fulfilled with other radiation therapy devices, the latter can be used for treatment as well. Organs-at-risk (rectal wall, bladder wall, bladder neck, urethra, as well as contralateral neurovascular bundles, contralateral external sphincter and contralateral pudendal vessels) are delineated (see constraints used in the first citation). Gross target volume (GTV) is delineated on the MRI while considering the hypointense T2-weighted nodule, the hypointense apparent diffusion coefficient, and the hyperintense perfusion zone. At first, the GTV is expanded by 1cm in all directions to generate the clinical target volume (CTV). The CTV is then cropped to the limits of the prostate. If the volume ratio CTV/Prostate is under 30%, the expansion margin of the GTV is increased progressively within the prostate by 0.1 cm increments so that the CTV achieves at least 30% of the prostate volume. Hence, a maximum of 1.5 cm margin around the GTV is allowed and encouraged. The CTV is then expanded by 3 mm to generate the planning target volume (PTV).

ELIGIBILITY:
* Inclusion Criteria (all the criteria must be fulfilled ) :

  * a. Localized prostate adenocarcinoma CAPRA score ≤ 5. This lesion is considered the Index lesion
  * b. Macroscopic tumor PIRADS score >4 on multiparametric MRI
  * c. The biopsies must be pathologic in or in the direct vicinity (the same prostatic zone defined as a quarter volume of the prostate (PZ)) of the MRI pathologic nodule
  * d. The absence of MRI pathologic criteria (PIRADS ≤3) in a Gleason score ≤ 6 (3+3)-ISUP Grade1 zone outside of the single Index lesion is considered clinically non-significant and does not preclude inclusion
  * e. The lesion can be plurifocal in a same intent to treat PZ
  * f. WHO Performance Status 0-1
  * g. No major urinary symptoms with IPSS score ≤15 and urinary continence ICIQ score =0
  * h. Patient is candidate for AS
* Exclusion Criteria :

  * a. Age at diagnosis < 50 years
  * b. Time between initial diagnostic biopsies and randomization > 4 months, or radiation therapy initiation > 6 months
  * c. Cribriform or Intraductal histologic components
  * d. Gleason Score ≥7 (3+4)-ISUP Grade 2 biopsy outside the intent to treat PZ
  * e. Multicentric pathologic MRI (PIRADS ≥4) outside a same PZ
  * f. Initial PSA > 20 ng/ml
  * g. Regional pathologic nodes or metastases
  * h. Androgen-deprivation therapy
  * i. Any cancer within the last 5 years except skin basocellular carcinoma or any uncontrolled cancer
  * j. Urethral stenosis
  * k. Recurrent prostatitis (at least 3 episodes within the last 3 years)
  * l. Any inflammatory collagen disease.
  * m. Contraindication to repeated prostatic biopsies or MRI

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
Rescue treatment performed or not | 5 years from the enrollment to the last follow up exams
  Rescue treatment performed due to:
  1. Recurrence - evolution (including at least one of these criteria) :
  1a. Any pathologic overscoring shift on biopsies examination
  1b. Any PSA doubling time < 9 months
  1c. Any doubling volume of the initial disease at MRI or appearance of a new prostatic lesion PIRADS ≥4
  1d. Regional or distant dissemination 2. Patient's personal decision or tumor board decision

SECONDARY OUTCOMES:
Clinical disease free survival | 5 years
  Parameter reporting any local, regional or distant disease recurrence
International Prostate Symptom Score (IPSS) | 5 years
  The score evaluates the quality of urinary fonction (score: 0-35). Higher score indicates worse outcome.
International Consultation on Incontinence Questionnaire (ICIQ). | 5 years
  The score evaluates urinary continence (score: 0-21). Higher score indicates worse outcome.
International Index of Erectile Function - 5 item version (IIEF5) | 5 years
  The index evaluates the quality of sexual founction (index: 5-25). Higher index indicates better function.
Hospital Anxiety and Depression Scale (HADS) | 5 years
  The scale evaluates anxiety and depression. Anxiety subscore(0-21). Depression subscore (0-21). An higher value indicates worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Nickers, MD, PhD, Principal Investigator — University Hospital Liège, Belgium; Mareva Lamande, MD, Principal Investigator — University Hospital Liège, Belgium
Locations (2):
- Belgium (2):
  - Vivalia Hospitals, Arlon
  - University Hospital Liège, Liège

IPD SHARING:
Plan to Share IPD: No
Forbidden according EU regulations. If Wished by researchers, they will have first to obtain the consent of the patients

REFERENCES:
- [Background] Nguyen PV, Donneaux B, Louis C, Bodgal Z, Philippi S, Biver S, Frederick B, Harze L, Lasar Y, Vogin G, Nickers P. Stereotactic focal radiotherapy as an alternative treatment for low-risk prostate cancer: Results of a single-arm monocenter Phase-II trial. Front Oncol. 2023 Apr 6;13:1143716. doi: 10.3389/fonc.2023.1143716. eCollection 2023. PMID 37091187
- [Background] Newcomb LF, Schenk JM, Zheng Y, Liu M, Zhu K, Brooks JD, Carroll PR, Dash A, de la Calle CM, Ellis WJ, Filson CP, Gleave ME, Liss MA, Martin F, McKenney JK, Morgan TM, Tretiakova MS, Wagner AA, Nelson PS, Lin DW. Long-Term Outcomes in Patients Using Protocol-Directed Active Surveillance for Prostate Cancer. JAMA. 2024 Jun 25;331(24):2084-2093. doi: 10.1001/jama.2024.6695. PMID 38814624
- [Background] Hopstaken JS, Bomers JGR, Sedelaar MJP, Valerio M, Futterer JJ, Rovers MM. An Updated Systematic Review on Focal Therapy in Localized Prostate Cancer: What Has Changed over the Past 5 Years? Eur Urol. 2022 Jan;81(1):5-33. doi: 10.1016/j.eururo.2021.08.005. Epub 2021 Sep 4. PMID 34489140
- [Background] Hamdy FC, Donovan JL, Lane JA, Metcalfe C, Davis M, Turner EL, Martin RM, Young GJ, Walsh EI, Bryant RJ, Bollina P, Doble A, Doherty A, Gillatt D, Gnanapragasam V, Hughes O, Kockelbergh R, Kynaston H, Paul A, Paez E, Powell P, Rosario DJ, Rowe E, Mason M, Catto JWF, Peters TJ, Oxley J, Williams NJ, Staffurth J, Neal DE; ProtecT Study Group. Fifteen-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Prostate Cancer. N Engl J Med. 2023 Apr 27;388(17):1547-1558. doi: 10.1056/NEJMoa2214122. Epub 2023 Mar 11. PMID 36912538